CLINICAL TRIAL: NCT05481619
Title: Changes in Intestinal Microecology Before and After Vedolizumab Treatment for Ulcerative Colitis and Correlation With Efficacy
Brief Title: Study of the Effect of Vedolizumab on Intestinal Microecological Changes and Its Efficacy in the Treatment of Ulcerative Colitis
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: I20210001091
Record Dates: First submitted 2022-07-25; First posted 2022-08-01 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — vedolizumab

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group of UC patients treated with vedolizumab (Active Comparator): Generic Name：vedolizumab Specification：300mg/bottle Dosage and Method of Administration：Usual adult dose for ulcerative colitis.300 mg IV every 30 minutes at weeks 0, 2, and 6, then every 8 weeks
  Interventions: Drug: Vedolizumab
- Normal control group (No Intervention): On the basis of the exclusion criteria, there are no significant intestinal inflammatory, autoimmune or neoplastic disorders.

INTERVENTIONS:
Drug: Vedolizumab — Recommended dose in patients with UC: 300 mg intravenously at weeks 0, 2, and 6 and every 8 weeks thereafter.
  Discontinue vedolizumab at week 14 in patients who do not show treatment benefit.
  Arms: Group of UC patients treated with vedolizumab

SUMMARY:
Inflammatory bowel disease is a group of chronic, non-specific inflammatory diseases of the intestinal tract whose etiology has not yet been fully elucidated, including ulcerative colitis and Crohn's disease. Vedolizumab, a novel biologic agent, is a recombinant humanized monoclonal antibody that specifically antagonizes intestine-selective α4β7 integrins on the surface of leukocyte subsets, thereby preventing migration of leukocyte subsets from the blood to the intestinal mucosa and reducing local inflammation in the gut. In this study the investigators propose to build on an existing cohort and analyse, by means of a multi-omics approach, the baseline gut microbial composition and abundance, intestinal and serum metabolome characteristics of UC patients and their changes during treatment, to predict the functional mechanisms by which these changing characteristics influence the therapeutic response to vindolizumab.

DETAILED DESCRIPTION:
Stool and blood samples etc. were taken from a cohort of patients with ulcerative colitis treated with Vedolizum at the Department of Gastroenterology, Second Affiliated Hospital of Zhejiang University School of Medicine as well as from a cohort of normal volunteers. Stool and blood samples from UC patients were analyzed at baseline and at 14, 30, and 52 weeks after starting treatment. Analysis of changes in gut microbial composition and abundance, gut and serum metabolome characteristics during 52 weeks of treatment in patients with UC. A model for predicting the efficacy of vedolizumab treatment by baseline gut microbial composition and abundance, and gut and serum metabolomic characteristics in patients with ulcerative colitis was developed in conjunction with clinical information from patients in the cohort. Based on the model developed, clinical and gut microbial composition and abundance, gut and serum metabolomics data from other UC patients published in public databases were combined to confirm the results already found using the UC cohort at our center.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older, with moderate to severe ulcerative colitis, with an indication for vedolizumab treatment;
2. Consent to participate in the study, read and sign the informed consent form;
3. No previous treatment with vedolizumab;
4. Never undergone biologic therapy or at least suspended previous biologic therapy for more than 12 weeks;
5. Not taking antibiotics or probiotics within the past 4 weeks.

Exclusion Criteria:

1. younger than 18 years of age;
2. pregnant or breastfeeding women;
3. patients who require the assistance of a surrogate, witness, or who are otherwise unable to complete the trial unaided;
4. other conditions that, in the opinion of the investigator, are unsuitable for enrollment or affect the subject's ability to complete the study;
5. have taken antibiotics or probiotics within the past 4 weeks;
6. have received prior treatment with vedolizumab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Remission rate of patients | 1 year
  Clinical remission response rates（Mayo score≤2）

SECONDARY OUTCOMES:
Baseline gut microbial composition and abundance of patients | 1 year
  Macro-genome sequencing of stool samples to analyze gut microbial composition and abundance
Gut and serum metabolome characteristics of UC patients | 1 year
  LC-MS mass spectrometry for faecal samples and serum samples to analyze metabolome characteristics

CONTACTS AND LOCATIONS:
Overall Officials: Yan Chen, Principal Investigator — 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China
Locations (1):
- Second Affiliated Hospital Zhejiang University School of Medicine, Zhengzhou, Hangzhou, China

IPD SHARING:
Plan to Share IPD: Yes
The results can be shared
Supporting Information: Study Protocol
Time Frame: now is available
Access Criteria: All the doctors